CLINICAL TRIAL: NCT00980590
Title: Airway Scope and Macintosh Laryngoscope for Tracheal Intubation in Patients Lying on the Ground
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 44-012
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2016-12

CONDITIONS: Intubation
Keywords: supine emergency intubations; emergency intubations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Airway Scope (Experimental): Intubation with Airway Scope
  Interventions: Device: Airway Scope
- Macintosh laryngoscope (Active Comparator): Intubation with Macintosh laryngoscope
  Interventions: Device: Macintosh Laryngoscope

INTERVENTIONS:
Device: Airway Scope — Tracheal intubation by Airway Scope
  Arms: Airway Scope
Device: Macintosh Laryngoscope — Tracheal intubation by Macintosh Laryngoscope
  Arms: Macintosh laryngoscope

SUMMARY:
Pre-hospital intubation is often required in sub-optimal conditions, such as in patients lying on the ground. Direct laryngoscopy and intubation of a patient lying supine on the ground is difficult because the intubator's head is far above the head of the patient. It is thus tricky to align the intubator's visual axis with the patient's tracheal axis. The Airway Scope is a new laryngoscope designed to facilitate intubation without requiring alignment of the oral, pharyngeal, and tracheal axes. We thus tested the hypothesis that the intubation with the Airway Scope is faster than the Macintosh laryngoscope in subjects lying on the ground.

DETAILED DESCRIPTION:
Adult surgical patients were enrolled. Following anesthesia induction and muscle relaxation, direct laryngoscopy was performed as usual and airway characteristics noted. Patients were randomly assigned to tracheal intubation by either the Airway Scope (n=50) or the Macintosh laryngoscope (n=50). Intubation was performed from a table positioned at the height as the operating table, thus simulating intubating on the ground. Overall intubation success rate, time required for intubation, the number of attempts required for successful intubation, and airway complications related to intubation were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for various surgeries requiring tracheal intubation as part of anesthesia and designated as American Society of Anesthesiologists (ASA) physical status I, II, or III.

Exclusion Criteria:

* Patients with an increased risk of pulmonary aspiration, cervical spine pathology, anticipated airway difficulties (i.e., Mallampati grade IV or thyromental distance <6 cm), and American Society of Anesthesiologists physical status >III.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Study Chair — The Cleveland Clinic; Ryu Komatsu, M.D., Principal Investigator — Kosei Hospital, Tokyo, Japan.
Locations (1):
- Kosei Hospital,., Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Airway Scope | Macintosh Laryngoscope
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Airway Scope | Macintosh Laryngoscope | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (19) | 53 (18) | 55 (20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 22 | 52
  Male | 20 | 28 | 48
Mouth opening [Mean (Standard Deviation); unit: cm] | 4.6 (0.7) | 4.7 (0.7) | 4.7 (0.7)
Height [Mean (Standard Deviation); unit: cm] | 158 (9) | 162 (9) | 160 (10)
Weight [Mean (Standard Deviation); unit: kg] | 56 (10) | 58 (10) | 57 (10)

OUTCOME MEASURES:

1. Primary Outcome: Intubation Time
Description: For the case with number of intubation attempt no more than 3, intubation time was defined as the total time of individual intubation attempt. Otherwise, intubation was defined as a failure and excluded from the calculation of intubation time.
Time Frame: The time from picking up the Airway Scope or Macintosh laryngoscope to confirmation of tracheal intubation by capnography.
Population: Patients with number of intubation attempt no more than 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Airway Scope | Macintosh Laryngoscope
Number analyzed (Participants) | 49 | 50
seconds | 18 (4) | 35 (16)

2. Secondary Outcome: Overall Intubation Success Rate
Time Frame: Intubation period
Measure: Number; unit: Percentage of overall intubation
Arm/Group | Airway Scope | Macintosh Laryngoscope
Number analyzed (Participants) | 50 | 50
Percentage of overall intubation | 98 | 100

3. Secondary Outcome: Number of Intubation Attempts
Time Frame: Intubation period
Measure: Number; unit: times
Arm/Group | Airway Scope | Macintosh Laryngoscope
Number analyzed (Participants) | 50 | 50
times
  1 | 37 | 45
  2 | 10 | 5
  3 | 3 | 0

4. Secondary Outcome: Incidence of Intubation Complications
Description: Including mucosal trauma, dental injury, lip injury, hypoxia (SPO2<95%) and Esophageal intubation
Time Frame: Intubation period
Measure: Number; unit: cases
Arm/Group | Airway Scope | Macintosh Laryngoscope
Number analyzed (Participants) | 50 | 50
cases
  Muscosal trauma | 2 | 5
  Dental injury | 0 | 1
  Lip injury | 4 | 6
  Hypoxia | 0 | 0
  Esophageal intubation | 0 | 1

ADVERSE EVENTS:
Arm/Group | Airway Scope | Macintosh Laryngoscope
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
Patients with anticipated airway difficulties were excluded. All intubations were performed by a single investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No